CLINICAL TRIAL: NCT00003928
Title: A Phase II Study Utilizing Gemcitabine and Cisplatinum in Patients With Renal Cell Carcinoma
Brief Title: Gemcitabine Plus Cisplatin in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3897; P30CA043703 (NIH); CWRU-3897; NCI-G99-1530
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin — Cisplatin IV over 60 minutes on day 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Drug: gemcitabine hydrochloride — Gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well gemcitabine and cisplatin work in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate of patients with metastatic renal cell carcinoma treated with gemcitabine and cisplatin.
* Assess toxicity of this regimen in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 60 minutes on day 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 4 months.

PROJECTED ACCRUAL: Approximately 29-38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic renal cell carcinoma
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Hematocrit at least 30%
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT no greater than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncontrolled hypertension
* No myocardial infarction within the past 8 weeks

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except nonmelanomatous skin cancer, carcinoma in situ of cervix, prostate intraepithelial neoplasia, or superficial bladder cancer
* No significant psychiatric disease
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 2 prior biologic response modifier regimens
* No concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed if measurable disease is outside radiation port
* At least 28 days since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Prior surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1999-01; Primary Completion 2005-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Assess the response rate of patients with metastatic renal cell carcinoma treated with gemcitabine and cisplatin. | Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States